CLINICAL TRIAL: NCT00535392
Title: Open-label, Single-arm, Multi-center, Pharmacokinetic, Safety and Tolerability Study of Levetiracetam Intravenous Infusion in Children (4 - 16 Years Old) With Epilepsy.
Brief Title: Open-label Study of Levetiracetam Intravenous Infusion in Children (4-16 Years Old) With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01274; 2006-005722-23 (EudraCT Number)
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-03

CONDITIONS: Epilepsy
Keywords: Epilepsy; Child; Levetiracetam; Keppra®; Infusion; Intravenous
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levetiracetam (Experimental)
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Intravenous 100 mg/mL, twice a day, maximum of 4 days
  Subjects on oral levetiracetam at study entry receive the same intravenous (IV) dosage (mg-for-mg) to their oral dose.
  Dosage for subjects not on levetiracetam at study entry was based on weight: if <50 kg, the dose was 20 mg/kg/day (10 mg/kg/day twice daily); if weight ≥ 50 kg, the dose of levetiracetam intravenous (LEV IV) was 1000 mg/day (500 mg twice daily).
  Other Names: ucb L059; Keppra®

SUMMARY:
Keppra injection is approved in the US as adjunctive therapy in the treatment of partial onset seizures in adults with epilepsy. The objective of the current study is to assess the safety, tolerability, and pharmacokinetics, of this formulation in children aged 4 to 16 years.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the safety and tolerability of levetiracetam intravenous 15-minute infusion administered every 12 hours, either as adjunctive treatment or monotherapy in children (4 to 16 years old) with epilepsy (except status epilepticus), either after switching from the equivalent levetiracetam oral dose administration or as a new antiepileptic treatment.

The evaluation period was to be considered as one complete set of 4 Pharmacokinetic (PK) samples for a maximum of 4 days;

* For children already taking levetiracetam oral tablets or oral solution prior to entering the study, the levetiracetam intravenous (LEV IV) dose will be equivalent (mg-for-mg) to their oral dose. The first intravenous (IV) infusion was to be administered 12 hours after the last oral dose of levetiracetam.
* For children not taking levetiracetam oral tablets or oral solution prior to entering the study:

  * If weight < 50 kg: dose of levetiracetam intravenous (LEV IV) dose will be calculated on the basis of their weight at 20 mg/kg/day (i.e. 10 mg/kg twice daily).
  * If weight ≥ 50 kg: dose of levetiracetam intravenous (LEV IV) will be 1000 mg/day (i.e. 500 mg twice daily).

However, when necessary for the safety of the subject or when the investigator deemed it appropriate the levetiracetam intravenous (LEV IV) dose could be modified after one day.

Subjects were hospitalized for the duration of the levetiracetam IV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 4 and 16 years of age, inclusive
* The subject suffers from epilepsy (except status epilepticus)
* The subject is requiring levetiracetam IV treatment in place of oral therapy for a short period of time

Exclusion Criteria:

* The subject has difficult venous accessibility
* History of status epilepticus during the 3 months prior to visit 1.
* The subject is taking felbamate at visit 1 or has been taking it in the past.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2007-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (25):
- United States (9):
  - La Jolla, California
  - Boston, Massachusetts
  - Chesterfield, Missouri
  - Buffalo, New York
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Richmond, Virginia
  - Milwaukee, Wisconsin
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- France (3):
  - Amiens
  - Lille
  - Paris
- Germany (2):
  - Heidelberg
  - Kehl
- Mexico (6):
  - Torreón, Coahuila
  - Puebla City, CP
  - Aguascalientes
  - Guadalajara
  - Mexico City
  - Puebla City
- Turkey (Türkiye) (2):
  - Ankara
  - Izmir

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from sites in the United States, Belgium, Germany, France, Mexico, and Turkey. The study began in September 2007 and continued until February 2010, with the last subject's visit occurring in February of 2010.
Period: Overall Study
Arm/Group | Levetiracetam
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Levetiracetam
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.71 (3.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Region of Enrollment [Number; unit: participants]
  France | 4
  United States | 7
  Mexico | 10
  Belgium | 5
  Turkey | 6
  Germany | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting at Least 1 Treatment-Emergent Adverse Event (TEAE) During the Treatment Period (up to 4 Days)
Time Frame: Treatment period (up to 4 days)
Population: All 33 subjects enrolled in the study were in the Intent to Treat (ITT) population and are included in this analysis.
Measure: Number; unit: Subjects
Arm/Group | Levetiracetam
Number analyzed (Participants) | 33
Subjects | 21

2. Secondary Outcome: Number of Subjects Who Received High-dose Levetiracetam Intravenous (LEV IV) (More Than 40 mg/kg/Day) During the Treatment Period (up to 4 Days)
Time Frame: Treatment period (up to 4 days)
Population: All 33 subjects enrolled in the study were in the Intent to Treat (ITT) population and are included in this analysis.
Measure: Number; unit: Subjects
Arm/Group | Levetiracetam
Number analyzed (Participants) | 33
Subjects | 10

3. Secondary Outcome: Number of Consecutive Levetiracetam Intravenous (LEV IV) Doses Received
Time Frame: Treatment period (up to 4 days)
Population: All 33 subjects enrolled in the study were in the Intent to Treat (ITT) population and are included in this analysis.
Measure: Mean (Standard Deviation); unit: Consecutive doses
Arm/Group | Levetiracetam
Number analyzed (Participants) | 33
Consecutive doses | 3.73 (1.61)

ADVERSE EVENTS:
Time Frame: Up to 4 days
Arm/Group | Levetiracetam
Serious Adverse Events (participants affected / at risk) | 3/33
Other Adverse Events (participants affected / at risk) | 12/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=33)
VOMITING (Gastrointestinal disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=33)
NAUSEA (Gastrointestinal disorders) | 3 (3)
DRY MOUTH (Gastrointestinal disorders) | 3 (3)
VOMITING (Gastrointestinal disorders) | 2 (3)
PYREXIA (General disorders) | 2 (3)
WEIGHT DECREASED (Investigations) | 2 (2)
CONVULSION (Nervous system disorders) | 3 (5)
SOMNOLENCE (Nervous system disorders) | 2 (7)
HYPOTENSION (Vascular disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.